CLINICAL TRIAL: NCT01280695
Title: A Phase 2a, Randomized, Double-Blind, Comparator- and Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability and Efficacy of Three Dose Levels of MSCD-0602 in Type 2 Diabetic Patients
Brief Title: A Randomized, Double-Blind, Comparator- and Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability and Efficacy of Three Dose Levels of MSDC-0602 in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metabolic Solutions Development Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSDC-0602-C002
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2; Diabetes Mellitus; Diabetes; High blood sugar; Blood sugar; Blood glucose; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia | interventions — MSDC-0602; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo capsule once daily
  Interventions: Drug: Placebo
- MSDC-0602 100 mg (Experimental): MSDC-0602 capsule 100 mg once daily
  Interventions: Drug: MSDC-0602 100 mg
- MSDC-0602 250 mg (Experimental): MSDC-0602 capsule 250 mg once daily
  Interventions: Drug: MSDC-0602 250 mg
- MSDC-0602 500 mg (Experimental): MSDC-0602 capsule 500 mg once daily
  Interventions: Drug: MSDC-0602 250 mg
- Pioglitazone 45 mg (Active Comparator): Pioglitazone capsule 45 mg once daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Placebo — Placebo Capsules
  Arms: Placebo
Drug: MSDC-0602 100 mg — MSDC-0602 100 mg Capsules
  Arms: MSDC-0602 100 mg
Drug: MSDC-0602 250 mg — MSDC-0602 250 mg Capsules
  Arms: MSDC-0602 250 mg
Drug: MSDC-0602 250 mg — MSDC-0602 500 mg Capsules
  Arms: MSDC-0602 500 mg
Drug: Pioglitazone — Pioglitazone 45 mg Capsules
  Arms: Pioglitazone 45 mg

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MSDC-0602 and to evaluate the reduction in fasting plasma glucose in patients with Type 2 diabetes.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

Inclusion Criteria:

1. Males and females with Type 2 diabetes (fasting plasma glucose ≥126 mg/dL at screening, glycosylated hemoglobin [HbA1c] >7 and ≤10%, and Insulin C-peptide >1 ng/mL). Patients can be naïve to diabetes therapy or if taking metformin should be on a stable dose level for a period of at least 3 months prior to screening visit (no dose limit).
2. Between the ages of 18-75 years, inclusive.
3. Females should be either postmenopausal (at least 12 months since last menses) or surgically sterilized (bilateral tubal ligation or hysterectomy). Menopausal status will be verified by a follicle-stimulating hormone (FSH) test. If FSH levels are below 40 mIU/mL, some method of birth control must be used. Those with bilateral tubal ligation must also use a barrier method of birth control. In addition, all females must have a negative pregnancy test at Screen and Day 15 regardless of childbearing potential. For postmenopausal women only, if FSH levels are above 40 mIU/mL and serum pregnancy results are indeterminant, the subject will be assessed as not pregnant.

   Males with female partners of child-bearing potential must agree to use adequate contraceptive methods (including a condom, plus one other form of contraception) if engaging in sexual intercourse.
4. Body Mass Index (BMI) ≥ 25 kg/m2 and ≤ 45 kg/m2 (inclusive).
5. Willing and able to make a screening visit to the clinic and six visits over a 10 week period.
6. Willing and able to sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.

Subject Exclusion Criteria:

1. Use of TZDs or diabetes medications other than metformin (generic or Glucophage®) 3 months prior to screening.
2. History of diabetic ketoacidosis or hyperosmolar non-ketotic coma.
3. Fasting plasma glucose in excess of 240 mg/dl at screening
4. History of heart failure (including CHF) or previous cardiovascular event (myocardial infarct, by-pass surgery, or PTCA) within the past 6 months prior to screening.
5. ALT and/or AST levels that equal or exceed twice the upper limit of normal; bilirubin levels that exceed 2 mg/dL; serum creatinine >1.5 mg/dL in men or > 1.4 mg/dL in women.
6. History of nephropathy, neuropathy, or retinopathy within 6 months of screening.
7. Use of glucocorticoids (oral, injectible, intraarticular, or chronic inhaled) or weight-loss drugs within 3 months of randomization.
8. Current or recurrent disease that may affect the action, absorption or disposition of the study treatment, or clinical or laboratory assessments.
9. Current or history of severe or unstable disorder (medical or psychiatric) requiring treatment that may make the patient unlikely to complete the study.
10. Febrile illness within the 5 days prior to Visit 1.
11. Known history of HIV, hepatitis B, or hepatitis C.
12. Clinically significant findings on physical examination, including BP, pulse rate and 12-lead ECG.
13. Blood pressure greater than 160/100 mmHg. Patients with elevated BP (<160/100 mmHg) with or without current treatment will be allowed at the discretion of the Principal Investigator (PI) and primary care physician. Individuals with hypertension must have been stabilized to the current treatment regimen for at least 6 weeks prior to screening.
14. Change in BP or lipid-lowering medication within 6 weeks or change in dose of metformin or thyroid replacement within 3 months prior to screening.
15. Known or suspected intolerance or hypersensitivity to the study drugs, closely related compounds or any of their stated ingredients.
16. History of alcohol or drug abuse within 6 months of Screening.
17. Have participated in an investigational study or received an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
18. Blood donation of 1 pint or more within 56 days of screening.
19. Plasmapheresis or plasma donation within 30 days of screening.
20. Single 12-lead ECG demonstrating a QTcB >450 msec at Screening. A single repeat ECG may be done at the Investigator's discretion.
21. Any surgical or medical condition which may significantly alter the absorption of any drug substance including, but not limited to, any of the following: history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling, or gastric banding, currently active inflammatory bowel syndrome.
22. Evidence of clinically relevant pathology that could interfere with the study results or put the patient's safety at risk.
23. Malignancy, including leukemia and lymphoma (not including basal cell skin cancer) within the last 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Colca, PhD, Study Director — Metabolic Solutions Development Company
Locations (14):
- United States (14):
  - Goodyear, Arizona
  - Chula Vista, California
  - Los Angeles, California
  - Bradenton, Florida
  - Hialeah, Florida
  - Pembroke Pines, Florida
  - Chicago, Illinois
  - Butte, Montana
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Charleston, South Carolina
  - Austin, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 investigational sites between February 15, 2011 and July 6, 2011.
Pre-assignment Details: This study consisted of a 14-day placebo lead-in period and a 28-day double-blind treatment period. Eligible patients were randomized following the lead-in period based on a stratification criterion of current metformin use (yes, no) to one of the 5 treatments: MSDC 0602 100 mg, MSDC-0602 250 mg, MSDC-0602 500 mg, pioglitazone 45 mg, or placebo.
Period: Overall Study
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Started | 26 | 25 | 26 | 26 | 26
Completed | 26 | 24 | 21 | 22 | 24
Not Completed | 0 | 1 | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg | Total
Number analyzed (Participants) | 26 | 25 | 26 | 26 | 26 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.87) | 57.6 (8.07) | 57.7 (7.35) | 55.5 (8.59) | 55.7 (8.01) | 56.7 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 13 | 10 | 14 | 52
  Male | 20 | 16 | 13 | 16 | 12 | 77
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 26 | 26 | 26 | 129

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: To characterize the reduction in fasting plasma glucose in response to three different doses of MSDC-0602 Tablets as compared to placebo following once-daily dosing for 28 consecutive days in patients with Type 2 diabetes.
Time Frame: Baseline and 28 days
Population: Per-Protocol Population:Included all patients who completed the 4-week, double blind treatment period without any major deviations from the protocol procedures. The Per-Protocol Population was used for all efficacy measurements.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 26 | 22 | 21 | 22 | 23
mg/dL | 6.0 (8.90) [-12.0 to 26.0] | -0.5 (9.77) [-34.0 to 19.0] | -20.0 (10.06) [-32.0 to 20.0] | -16.0 (9.68) [-37.0 to 10.0] | -22.0 (9.38) [-47.0 to -4.0]
Statistical Analysis 1: Comparison: Placebo vs MSDC-0602 100 mg; Test type: Superiority or Other; p = 0.4195, Wilcoxon (Mann-Whitney); Median Difference (Net) = -10.0, 95% CI 2-sided [-34.0 to 14.0]
Statistical Analysis 2: Comparison: Placebo vs MSDC-0602 250 mg; Test type: Superiority or Other; p = 0.0811, Wilcoxon (Mann-Whitney); Median Difference (Net) = -18.0, 95% CI 2-sided [-38.0 to 4.0]
Statistical Analysis 3: Comparison: Placebo vs MSDC-0602 500 mg; Test type: Superiority or Other; p = 0.0639, Wilcoxon (Mann-Whitney); Median Difference (Net) = -20.0, 95% CI 2-sided [-38.0 to 1.0]
Statistical Analysis 4: Comparison: Placebo vs Pioglitazone 45 mg; Test type: Superiority or Other; p = 0.0022, Wilcoxon (Mann-Whitney); Median Difference (Net) = -32.0, 95% CI 2-sided [-50.0 to -12.0]

2. Secondary Outcome: Change From Baseline in HbA1c
Description: To explore the drug effect difference in the reduction in hemoglobin A1c in response to three different doses of MSDC-0602 and pioglitazone (45 mg Actos®) as compared to placebo following once-daily dosing for 28 consecutive days in patients with Type 2 diabetes.
Time Frame: Baseline and 28 days
Population: The Per-Protocol Population included all patients who completed the 4-week, double blind treatment period without any major deviations from the protocol procedures.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 26 | 22 | 21 | 22 | 23
percentage of hemoglobin | 0.14 (0.081) | 0.09 (0.088) | -0.10 (0.090) | -0.17 (0.088) | -0.14 (0.086)

3. Secondary Outcome: Change From Baseline in Body Weight
Description: To characterize the effects of three different doses of MSDC-0602 and pioglitazone as compared to placebo on hematocrit, body weight, and edema following once-daily dosing for 28 consecutive days in patients with Type 2 diabetes.
Time Frame: Baseline and 28 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 26 | 22 | 21 | 22 | 23
kg | 0.12 (0.267) | 0.25 (0.291) | -0.07 (0.297) | 0.17 (0.290) | 0.54 (0.284)

4. Secondary Outcome: Change From Baseline in Hematocrit
Description: To characterize the effects of three different doses of MSDC-0602 and pioglitazone as compared to placebo in hematocrit following once-daily dosing for 28 consecutive days in patients with Type 2 diabetes.
Time Frame: Baseline and 28 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Change from baseline
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 26 | 22 | 21 | 22 | 23
Change from baseline | -0.9 (0.36) | -0.9 (0.39) | -1.2 (0.40) | -1.7 (0.39) | -1.4 (0.38)

5. Secondary Outcome: Change in Fasting Plasma Insulin
Description: To characterize the effects of 3 different doses of MSDC-0602 and pioglitazone as compared to placebo on insulin following once-daily dosing for 28 consecutive days
Time Frame: Baseline and 28 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 26 | 22 | 21 | 22 | 23
µIU/mL | 3.06 (1.434) | -1.70 (1.561) | -1.11 (1.601) | -2.13 (1.564) | -3.21 (1.523)

6. Secondary Outcome: Change From Baseline in High Molecular Weight Adiponectin
Description: To evaluate the effects of three different doses of MSDC-0602 and pioglitazone as compared to placebo on biomarkers of inflammatory status (high molecular weight adiponectin) following once-daily dosing for 28 consecutive days in patients with Type 2 diabetes.
Time Frame: Baseline and 28 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 26 | 22 | 21 | 22 | 23
ng/mL | 3.6 (15.28) | 44.1 (17.30) | 101.6 (17.00) | 139.2 (16.62) | 206.0 (16.35)

ADVERSE EVENTS:
Arm/Group | Placebo | MSDC-0602 100 mg | MSDC-0602 250 mg | MSDC-0602 500 mg | Pioglitazone 45 mg
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 2/26 | 0/25 | 1/26 | 5/26 | 4/26
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=26) | MSDC-0602 100 mg (N=25) | MSDC-0602 250 mg (N=26) | MSDC-0602 500 mg (N=26) | Pioglitazone 45 mg (N=26)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0/25 (0) | 2 (2)
Edema peripheral (General disorders) | 2 (2) | 0 (0) | 0/25 (0) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less